CLINICAL TRIAL: NCT07372638
Title: Sensorised Surgical Gloves for Neuroendovascular Procedures: Preclinical Study in Flow Diverter Placement Using 3D Printed Biorealistic Haptic Simulators
Brief Title: Sensorised Surgical Gloves for Neuroendovascular Procedures
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: R&D No. 2025/0166; REC No. 25/NS/0083 (Other: North of Scotland Research Ethics Committee (1)); IRAS Project ID 331897 (Other: NHS Health Research Authority)
Record Dates: First submitted 2025-11-19; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Endovascular Procedures; Force Sensing Surgical Gloves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Simulated FD procedure (Experimental)
  Interventions: Device: Sensorised surgical gloves; Device: Computer vision

INTERVENTIONS:
Device: Sensorised surgical gloves — Force sensing surgical gloves
Device: Computer vision — Data collection to investigate potential for computer vision

SUMMARY:
A deeper understanding of the forces required for optimal flow diverter stent deployment could improve procedural safety and shorten the learning curve for new devices. In the past, force sensors have been physically attached to devices in some way. The investigators approach is to incorporate force sensors into the hands of the operator handling the device using sensorised surgical gloves. Participants will be asked to deploy a Flow Diverter (FD) in a biorealistic silicone model while wearing force sensing surgical gloves. The primary objective of the study is to show whether sensorised gloves are capable of meaningful force detection in neurointerventional procedures. The investigators will also explore the potential of developing computer vision technology in neurointervention. The investigators are inviting groups of experts and novices to participate. This will allow the investigators to understand if analysis of glove force outputs can distinguish operator experience.

DETAILED DESCRIPTION:
Custom-made conducting melamine foam-based soft piezoresistive sensors will be fabricated and mounted on surgical gloves. Calibration and recording during testing will be made by measuring change in voltage. Participants will be asked to deploy a Pipeline Embolisation Device (Medtronic) in a silicone model. Continuous force recordings will be made, with measurement of the range of forces applied (N) during the procedure. The investigators will compare force recordings for expert and novice operators. Participants will be blinded to the forces they exert. Videos and fluoroscopy images will be recorded and objective structured assessment of technical skills (OSATS) performed.

ELIGIBILITY:
Inclusion Criteria:

- Experienced neurointerventionist or doctor in training.

Exclusion Criteria:

- No training in use of medical ionising radiation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Force detection from sensorised surgical gloves | Intra procedural
  Force (newtons) during flow diverter placement in a cerebral aneurysm model

SECONDARY OUTCOMES:
Objective structured assessment of technical skill (OSATS) | Intra procedural
  OSATS to evaluate task performance

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan J Downer, MRCP FRCR, Principal Investigator — NHS Lothian
Locations (1):
- Royal Infirmary of Edinburgh, Edinburgh, Scotland, United Kingdom